CLINICAL TRIAL: NCT06914284
Title: Apathy-related Neurobehavioral Markers of Cognitive Decline in Old-age Bipolar Disorders: Proof-of-concept
Acronym: ANACONDA
Status: Recruiting | Type: Observational
Sponsor: Hospital Center Guillaume Régnier (Other)
Collaborators: Rennes University Hospital (Other); Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_01_GR/ANACONDA; ID-RCB (Other: 2024-A00407-40)
Record Dates: First submitted 2024-09-03; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Apathy; Bipolar Disorder
Keywords: Apathy; Actimetry; Neurobehavioral marker; Cognitive decline; Old Age Bipolar Disorder; MRI; Speech marker
MeSH Terms: conditions — Lethargy; Bipolar Disorder; Cognitive Dysfunction | interventions — Actigraphy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Old Age Bipolar Disorder: the strategy procedure will consist of using actigraphy and MRI.
  The wGT3X-BT actigraph (wGT3x-BT) will be worn on the wrist for 5 days. The set up is made at Day 1. The actigraph will be programmed to automatically switch off after 4 full days of use (96 hours). After 5 full days (120 hours), the participant returns to the research center so the data are downloaded on a secured computer dedicated to store and analyse the data. At day 5, a MRI will be perform.The total acquisition time is about 45 minutes:
  * Degenerative: anatomical 3DT1 (~5 minutes acquisition).
  * Inflammation: multicompartment imaging models (~15 minutes acquisition) such as the Neurite Orientation and Dispersion Index (NODDI) are used to quantify in-vivo microstructure inflammation.
  * Vascular: 3D Fluid-attenuated inversion recovery (FLAIR ~5 minutes acquisition) and Arterial Spin labelling (ASL, ~8 minutes acquisition)
  * Functional connectivity: rs BOLD (~10 minutes acquisition)
  Interventions: Other: Actigraphy and MRI
- Healthy Controls: the strategy procedure will consist of using actigraphy and MRI.
  The wGT3X-BT actigraph (wGT3x-BT) will be worn on the wrist for 5 days. The set up is made at Day 1. The actigraph will be programmed to automatically switch off after 4 full days of use (96 hours). After 5 full days (120 hours), the participant returns to the research center so the data are downloaded on a secured computer dedicated to store and analyse the data. At day 5, a MRI will be perform.The total acquisition time is about 45 minutes:
  * Degenerative: anatomical 3DT1 (~5 minutes acquisition).
  * Inflammation: multicompartment imaging models (~15 minutes acquisition) such as the Neurite Orientation and Dispersion Index (NODDI) are used to quantify in-vivo microstructure inflammation.
  * Vascular: 3D Fluid-attenuated inversion recovery (FLAIR ~5 minutes acquisition) and Arterial Spin labelling (ASL, ~8 minutes acquisition)
  * Functional connectivity: rs BOLD (~10 minutes acquisition)
  Interventions: Other: Actigraphy and MRI

INTERVENTIONS:
Other: Actigraphy and MRI — All participants will wear a wGT3X-BT actigraph (wGT3x-BT) for 4 days. Actigraphs are collected back at Day 4, after full 96 hours, when coming to the MRI platform. There, they will undergo 45 minutes MRI that acquire MRI signals to quantify degenerative, inflammatory, vascular and functional cerebral features.

SUMMARY:
The goal of this clinical trial is to identify reliable markers of apathy in elderly subjects with bipolar disorder, age between 70 and 85 years, in order to accurately identify subjects at high risk of progressing to dementia by measuring motor activity (actimetrics), recorded language and analysing brain changes (MRI).

Actimetry is the measurement and recording of body movements using an actimeter. This device is worn on the wrist and contains sensors capable of measuring and recording all movements, including those of very low intensity. An automated speech analysis using artificial intelligence is used to detect low-intensity anomalies, and we want to test whether individual differences correspond to individual differences in brain anatomy and function.

Researchers will compare elderly subjects with bipolar disorder and healthy volunteer, age between 70 and 85 years.

Participants will be asked to:

* Perform an MRI
* Complete 3 cognitive tests: verbal memory, verbal fluency and an emotional storytelling task, in which you will be asked to describe a memory orally using positive, negative and neutral emotions.
* wear an actimeter on your wrist for 4 days.

ELIGIBILITY:
Inclusion Criteria:

1. Population: Age between 70 and 85 years-old, living at home (Participants living in nursing homes are not included).
2. Condition: OABD type 1, type 2 and type 3 assessed by the DSM5 criteria
3. Stable: no MDE or hypomanic state within the last 6 months
4. Ambulatory setting only
5. General condition: Successful Gait speed test from the Short Physical Performance Battery (SPPB): beingable to walk 4 meters in 4 seconds (SPPB NIH Toolbox)44
6. Person affiliated to a social security regime
7. Patients who have given their free, informed and written consent to take part in the study

Exclusion Criteria:

1. Psychiatric conditions and or co-morbidities

   1. Unipolar depression
   2. Recurrent unipolar depression
   3. Substance use disorder according to DSM5 criteria. Benzodiaepine and/or z-drugs dependence are accepted.
2. Neurological and cerebral co-morbidities

   1. Major Cognitive Disorder: significant cognitive decline characterized by extensive cognitive tests or at least a standardized clinical evaluation AND at least loss of autonomy in complex instrumental daily living function, not related to delirium (DSM5 criteria)
   2. Medical history of known degenerative disorders: Alzheimer's disease, Lobar Degenerative Fronto-temporal disorders, Lewy Body disease, corticobasal degenerative disorder, Supranuclear Palsy, epilepsy.
   3. Medical history of known Parkinson's disease (according to the Movement Disorder Society (MDS)45 criteria)
   4. Medical history of known stroke
   5. Severe Parkinsonism (defined by MDS-Unified Parkinson's Disease Rating Scale46 > 20)
3. MRI contra-indications: metallic implants, severe claustrophobia
4. Adults under legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty.
5. Hospitalized at inclusion

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients treated in the old-age psychiatry department of the Pôle Hospitalo-Universitaire de Psychiatrie Adulte (PHUPA) for OABD may be offered participation in the study. Eligible patients according to the inclusion criteria will be recruited during standard visits at CHGR. Informed consent along with a document describing the study will be presented during visit.
  Healthy volunteers will be recruited from the patient's relatives and/or via posters and/or the CHGR's internal networks.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Compare Actigraphic measures acquired by OABD participants and with those of Healthy controls (HC) | during 4 days
  These very complex and highly dimensional signals are reduced to a sum, for a given period of time, of the variations in acceleration (in g/sec) after pre-processing (band-pass filtering) for each participants (OABD and healthy controls

SECONDARY OUTCOMES:
speech biomarkers :Temporal, Source, Prosodic and Spectral speech features automatically derived from the audio recordings of 3 cognitive tasks. | baseline and only for OABD participants at 12 month and 36 month
  To identify a set of speech biomarkers, specific to OABD (compared to HC), 3 cognitive tasks , verbal learning (with the Rey Auditory Verbal Learning Task), semantic verbal fluency task and narrative storytelling are implemented on the Milli® platform. Each of these tasks enable to derive temporal, source, prosodic and spectral features from remote recordings.
MRI derived cerebral features, specific to OABD participants compared to Healthy control | at Day 4
  measure cortical thickness and sub-cortical volumes to identify degenerative alterations measure water diffusion in several cellular compartments and appropriate multi compartment modeling (MCM) such as Neurite Orientation Diffusion and Dispersion Index (NODDI) to identify Inflammation Measure tissue blood flow Using arterial spin labeling (ASL) to identify Vascular health

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel RG ROBERT, Principal Investigator — HC Guillaume Regnier
Locations (1):
- Centre Hospitalier Guillaume Regnier, Rennes, Ile Et Vilaine, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu YT, Beiser AS, Breteler MMB, Fratiglioni L, Helmer C, Hendrie HC, Honda H, Ikram MA, Langa KM, Lobo A, Matthews FE, Ohara T, Peres K, Qiu C, Seshadri S, Sjolund BM, Skoog I, Brayne C. The changing prevalence and incidence of dementia over time - current evidence. Nat Rev Neurol. 2017 Jun;13(6):327-339. doi: 10.1038/nrneurol.2017.63. Epub 2017 May 12. PMID 28497805
- [Background] Richmond-Rakerd LS, D'Souza S, Milne BJ, Caspi A, Moffitt TE. Longitudinal Associations of Mental Disorders With Dementia: 30-Year Analysis of 1.7 Million New Zealand Citizens. JAMA Psychiatry. 2022 Apr 1;79(4):333-340. doi: 10.1001/jamapsychiatry.2021.4377. PMID 35171209
- [Background] Diniz BS, Butters MA, Albert SM, Dew MA, Reynolds CF 3rd. Late-life depression and risk of vascular dementia and Alzheimer's disease: systematic review and meta-analysis of community-based cohort studies. Br J Psychiatry. 2013 May;202(5):329-35. doi: 10.1192/bjp.bp.112.118307. PMID 23637108
- [Background] Byers AL, Yaffe K. Depression and risk of developing dementia. Nat Rev Neurol. 2011 May 3;7(6):323-31. doi: 10.1038/nrneurol.2011.60. PMID 21537355
- [Background] Wu JJ, Wang HX, Yao W, Yan Z, Pei JJ. Late-life depression and the risk of dementia in 14 countries: a 10-year follow-up study from the Survey of Health, Ageing and Retirement in Europe. J Affect Disord. 2020 Sep 1;274:671-677. doi: 10.1016/j.jad.2020.05.059. Epub 2020 May 26. PMID 32664001
- [Background] Kaup AR, Byers AL, Falvey C, Simonsick EM, Satterfield S, Ayonayon HN, Smagula SF, Rubin SM, Yaffe K. Trajectories of Depressive Symptoms in Older Adults and Risk of Dementia. JAMA Psychiatry. 2016 May 1;73(5):525-31. doi: 10.1001/jamapsychiatry.2016.0004. PMID 26982217
- [Background] Almeida OP, McCaul K, Hankey GJ, Yeap BB, Golledge J, Flicker L. Risk of dementia and death in community-dwelling older men with bipolar disorder. Br J Psychiatry. 2016 Aug;209(2):121-6. doi: 10.1192/bjp.bp.115.180059. Epub 2016 Jun 9. PMID 27482038
- [Background] Velosa J, Delgado A, Finger E, Berk M, Kapczinski F, de Azevedo Cardoso T. Risk of dementia in bipolar disorder and the interplay of lithium: a systematic review and meta-analyses. Acta Psychiatr Scand. 2020 Jun;141(6):510-521. doi: 10.1111/acps.13153. Epub 2020 Feb 11. PMID 31954065
- [Background] Almeida OP, Hankey GJ, Yeap BB, Golledge J, Flicker L. Older men with bipolar disorder: Clinical associations with early and late onset illness. Int J Geriatr Psychiatry. 2018 Dec;33(12):1613-1619. doi: 10.1002/gps.4957. Epub 2018 Jul 17. PMID 30015397
- [Background] John A, Saunders R, Desai R, Bell G, Fearn C, Buckman JEJ, Brown B, Nurock S, Michael S, Ware P, Marchant NL, Aguirre E, Rio M, Cooper C, Pilling S, Richards M, Stott J. Associations between psychological therapy outcomes for depression and incidence of dementia. Psychol Med. 2023 Aug;53(11):4869-4879. doi: 10.1017/S0033291722002537. Epub 2022 Sep 15. PMID 36106698
- [Background] Stott J, Saunders R, Desai R, Bell G, Fearn C, Buckman JEJ, Brown B, Nurock S, Michael S, Ware P, Marchant NL, Aguirre E, Rio M, Cooper C, Pilling S, Richards M, John A. Associations between psychological intervention for anxiety disorders and risk of dementia: a prospective cohort study using national health-care records data in England. Lancet Healthy Longev. 2023 Jan;4(1):e12-e22. doi: 10.1016/S2666-7568(22)00242-2. Epub 2022 Dec 9. PMID 36509102
- [Background] Alexopoulos GS. Depression in the elderly. Lancet. 2005 Jun 4-10;365(9475):1961-70. doi: 10.1016/S0140-6736(05)66665-2. PMID 15936426
- [Background] van Dalen JW, van Wanrooij LL, Moll van Charante EP, Brayne C, van Gool WA, Richard E. Association of Apathy With Risk of Incident Dementia: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2018 Oct 1;75(10):1012-1021. doi: 10.1001/jamapsychiatry.2018.1877. PMID 30027214
- [Background] Ruthirakuhan M, Herrmann N, Vieira D, Gallagher D, Lanctot KL. The Roles of Apathy and Depression in Predicting Alzheimer Disease: A Longitudinal Analysis in Older Adults With Mild Cognitive Impairment. Am J Geriatr Psychiatry. 2019 Aug;27(8):873-882. doi: 10.1016/j.jagp.2019.02.003. Epub 2019 Feb 7. PMID 30910421
- [Background] Dujardin K, Sockeel P, Delliaux M, Destee A, Defebvre L. Apathy may herald cognitive decline and dementia in Parkinson's disease. Mov Disord. 2009 Dec 15;24(16):2391-7. doi: 10.1002/mds.22843. PMID 19908317